CLINICAL TRIAL: NCT07360288
Title: A Multi-center, Single-arm, Open-label Phase II Study to Evaluate the Efficacy and Safety of TC011 in Patients With Relapsed or Refractory Follicular Lymphoma
Brief Title: Efficacy and Safety of TC011 in Relapsed or Refractory Follicular Lymphoma
Acronym: TC011_FL_201
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: TICAROS Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TC011_FL_201
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Follicular Lymphoma (FL)
Keywords: Follicular Lymphoma; CAR-T; CD19; Adoptive Cell Therapy; Immunotherapy
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TC011 single-arm (Experimental): Single-arm, open-label study receiving TC011 infusion.
  Interventions: Biological: TC011 single-arm

INTERVENTIONS:
Biological: TC011 single-arm — CD19-targeted chimeric antigen receptor T-cell therapy

SUMMARY:
This Phase II, multi-center, single-arm, open-label study evaluates the efficacy and safety of TC011, a CD19-targeted CAR-T cell therapy, in adult patients with relapsed or refractory follicular lymphoma (Grade 1, 2, or 3a).

The primary endpoint is objective response rate (ORR) assessed by independent review using the Lugano 2014 classification.

DETAILED DESCRIPTION:
This is a multi-center, single-arm, open-label Phase II clinical trial designed to evaluate the efficacy and safety of TC011, a CD19-targeted chimeric antigen receptor T-cell (CAR-T) therapy, in adult patients with relapsed or refractory follicular lymphoma.

Eligible patients who meet all inclusion and exclusion criteria will undergo leukapheresis for the manufacture of TC011, followed by lymphodepleting chemotherapy and a single intravenous infusion of TC011. Patients will be followed according to the study schedule to assess efficacy and safety outcomes.

The primary efficacy endpoint is objective response rate assessed by independent review using standardized response criteria. Secondary endpoints include additional efficacy measures and safety evaluations. Exploratory assessments may include characterization of TC011-related cellular kinetics and biomarker analyses.

An independent Data Safety Monitoring Board will periodically review accumulated safety and efficacy data to ensure patient safety throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide written informed consent.
2. Age ≥19 years at the time of screening.
3. Histologically confirmed follicular lymphoma Grade 1, 2, or 3a according to WHO 2017 classification.
4. Relapsed or refractory disease after at least two prior systemic therapies including rituximab.
5. ECOG performance status ≤2.
6. Life expectancy ≥12 weeks.
7. At least one measurable lesion (long diameter ≥1.5 cm).
8. Adequate hepatic, renal, hematologic, pulmonary, and cardiac function.
9. Eligible for leukapheresis and successful manufacture of TC011.
10. Agreement to use effective contraception for at least 6 months after TC011 infusion.

Exclusion Criteria:

1. Histologic transformation to diffuse large B-cell lymphoma or follicular lymphoma Grade 3b.
2. Unresolved ≥Grade 2 toxicity from prior anticancer therapy (excluding hematologic abnormalities).
3. Active or prior malignancy within 2 years, except adequately treated non-melanoma skin cancer or carcinoma in situ.
4. Clinically significant cardiovascular disease within 6 months prior to screening.
5. Active central nervous system involvement by lymphoma.
6. Active uncontrolled infection, including HBV, HCV, HIV, or syphilis (protocol-defined exceptions apply).
7. Active autoimmune or inflammatory neurologic disease.
8. Rapidly progressive disease requiring urgent therapy.
9. Prior treatment with anti-CD19 therapy, adoptive T-cell therapy, gene therapy, or allogeneic stem cell transplantation.
10. Major surgery within 4 weeks prior to screening.
11. Use of investigational agents within 4 weeks prior to screening.
12. Known hypersensitivity to components of TC011.
13. Pregnant or breastfeeding women.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-05-31 (Estimated); Study Completion 2030-02-28 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 96 weeks
  Proportion of patients achieving CR or PR per 2014 Lugano classification by independent review

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to 96 weeks
  Proportion of subjects achieving complete response per 2014 Lugano classification by independent review
Disease Control Rate (DCR) | Up to 96 weeks
  Proportion of subjects with complete response, partial response, or stable disease
Stable Disease Rate (SDR) | Up to 96 weeks
  Proportion of subjects with stable disease per 2014 Lugano classification
Duration of Response (DOR) | Up to 96 weeks
  Time from first documentation of response (CR or PR) to disease progression or death from any cause
Time to Response (TTR) | Up to 96 weeks
  Time from TC011 infusion to first documented response (CR or PR)
Progression-Free Survival (PFS) | Up to 96 weeks
  Time from TC011 infusion to disease progression or death from any cause
Overall Survival (OS) | Up to 96 weeks
  Time from TC011 infusion to death from any cause
Incidence and severity of adverse events | Up to 96 weeks
  Incidence, severity, and type of adverse events graded per CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Won Seok Kim, MD, PhD, Principal Investigator — Samsung Medical Center, Department of Hematology-Oncology

IPD SHARING:
Plan to Share IPD: No